CLINICAL TRIAL: NCT04721288
Title: REmote moBile Outpatient mOnitoring in Transplant (Reboot) 2.0
Brief Title: REmote moBile Outpatient mOnitoring in Transplant 2.0
Acronym: Reboot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Heather Ross, Head, Division of Cardiology, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20-6082
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Solid Organ Transplant; Heart Transplant; Liver Transplant; Kidney Transplant
Keywords: mobile health; telemonitoring; transplantation; wearable sensors; solid organ transplant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 1 year of tailored communication with transplant care team through Reboot application in addition to standard of care communication system.
  Interventions: Other: Active communication through Reboot application
- Standard of Care Group (Sham Comparator): 1 year of generic communication through Reboot application with communication with transplant care team through standard of care communication system.
  Interventions: Other: Generic communication through Reboot application

INTERVENTIONS:
Other: Active communication through Reboot application — Access to active communication with the transplant care team through Reboot application based asynchronous messaging for non-urgent issues, as well as personalized clinical notifications.
  Arms: Intervention Group
Other: Generic communication through Reboot application — Access to generic messaging through Reboot application, and communication with the transplant care team through standard of care communication system.
  Arms: Standard of Care Group

SUMMARY:
This study is designed to determine if an innovative mobile health intervention designed to improve patient-provider communication can reduce unscheduled hospitalizations, and visits to the emergency department and ambulatory clinic in adult heart, liver, and kidney transplant patients.

DETAILED DESCRIPTION:
Mobile health technologies such as smartphones and wearable devices can remotely monitor health. These technologies hold promise to improve health outcomes in a spectrum of patients by providing health care teams with better connectivity which may prompt more timely responses to questions and improvements to care.

The purpose of this study is to evaluate if solid organ transplant (SOT) recipients benefit from improved monitoring and removal of communication barriers as the most common reasons for readmission and mortality may be mitigated by clinical intervention. Additionally, medication adherence is critical in transplant patients to prevent graft rejection. We anticipate that remote monitoring will improve medication adherence/adjustments, and will allow for identification of early health issues, reducing preventable hospital readmissions. Thus, this study will determine if an innovative mobile health intervention, designed to improve patient-clinician communication, reduces unnecessary hospital readmission and visits to the emergency department and transplant clinic when utilized in addition to the standard of care telephone communication system. We will also incorporate clinical and continuous ambulatory physiologic data collected as part of the mobile health intervention to develop machine learning algorithms capable of identifying early indicators of adverse outcomes in adult heart, kidney, and liver transplant patients.

We hypothesize that: the delivery of personalized communication using a mobile health application will improve patient self-management resulting in a 50% reduction in preventable hospital readmission, and unscheduled visits to the emergency department and transplant clinic. With tailored communication through the mobile health application, we expect fewer standard of care phone messages for patients in the intervention group and patients with higher activity levels (average daily step-count) pre-transplantation will have lower index hospitalization length of stay. Finally, the large dataset collected from this study will allow novel machine learning-derived risk prediction models to more accurately predict adverse outcomes (e.g., organ rejection, infection, and death), compared to conventional regression models.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ (heart, liver, or kidney) transplant patients
* The ability to use a smartphone
* English speaking

Exclusion Criteria:

* Poor health literacy (reading level less than grade 5)
* Inability to follow instructions from the Reboot application
* Transfer to a non-University Health Network Hospital for follow-up and management

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Unscheduled hospital admission or visit to emergency department or transplant clinic. | 1-month
  A composite score of unscheduled hospital admission, visit to the emergency department or ambulatory transplant clinic (i.e., total number of visits) will be calculated for each group at the pre-specified time intervals. A central adjudication committee will assess each readmission and visit to determine if they constitute a study event.

SECONDARY OUTCOMES:
EuroQol-5 (EQ-5D) Dimension questionnaire | 1-month, 3-months, 12-months
  The EQ-5D is a comprehensive and compact health status classification and health state preference questionnaire, widely used in many patient populations.
Patient-Reported Outcomes Measurement Information System (PROMIS) tool | 1-month, 3-months, 12-months
  PROMIS is a single patient-centered questionnaire that measures and monitors several domains, including physical, mental, and social health. It is validated for use with the general population and individuals living with chronic disease.
Graft survival rate | 12-months
  Transplanted organ survival rate will be calculated for each group at the end of the study period.
Patient survival rate | 12-months
  Patient survival rate will be calculated for each group at the end of the study period.
Easy Call interactions | 1-month, 3-months, 12-months
  The number of interactions that each group has with standard of care communication system ('Easy Call') will be compared.
Index hospitalization length of stay | 1-month
  Participants activity level while on the transplant waiting list will be quantified by their average daily step count, and compared to the length of their index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Heather Ross, MD, Principal Investigator — University Health Network, Toronto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murray KR, Foroutan F, Amadio JM, Posada JD, Kozuszko S, Duhamel J, Tsang K, Farkouh ME, McDonald M, Billia F, Barber E, Hershman SG, Bhat M, Tinckam KJ, Ross HJ, McIntosh C, Moayedi Y. Remote Mobile Outpatient Monitoring in Transplant (Reboot) 2.0: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2021 Oct 22;10(10):e26816. doi: 10.2196/26816. PMID 34528885